CLINICAL TRIAL: NCT04346927
Title: Investigation of the Effects of Exercise Using Telerehabilitation in Patients Diagnosed With Coronavirus (COVID-19) and Followed at Home
Brief Title: Telerehabilitation for Patients Diagnosed With Coronavirus
Acronym: COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yasemin Çırak (Other)
Responsible Party: Sponsor-Investigator, Yasemin Çırak, Physiotherapist, PhD, Associate Professor, Istinye University
Organization: Istinye University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 009
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Telerehabilitation; Coronavirus
Keywords: Exercise; Breathing exercise; physiotherapy
MeSH Terms: conditions — Coronavirus Infections; Motor Activity | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): The group to which the exercise protocol consisting of breathing exercises, posture exercises, peripheral muscle training and light aerobic exercises will be applied.
  Interventions: Other: Telerehabilitation
- Control Group (Active Comparator): group to be given an exercise brochure
  Interventions: Other: exercise brochure

INTERVENTIONS:
Other: Telerehabilitation — 15 volunteers diagnosed with coronavirus will be included in experimental group. An online exercise program has been created for individuals who will participate in the study. This program is planned to continue 3-4 days a week, in a 30-minute session and for 6 weeks. Treatment sessions will include breathing exercises, posture exercises, peripheral muscle exercises and light aerobic exercises. Individuals were asked to participate in the research via telerehabilitation connection system and were told that they would do their exercises with a physiotherapist.
  Arms: Study Group
Other: exercise brochure — 15 volunteers diagnosed with coronavirus will be included in control group.The same exercises will be given to the control group as a brochure and they will be asked to do it for 6 weeks.
  Arms: Control Group

SUMMARY:
In December 2019, new coronavirus pneumonia (COVID-19) erupted in Wuhan (Hubei, China) and quickly spread from a single city to the entire country. It did not take long for this epidemic to spread to the world. After that, World Health Organization declared this epidemic disease as a pandemic. As of now, the number of coronavirus deaths increased to 108,281 worldwide. Total number of cases approached 1,800,000 according to the latest information. While the number of healed patients was highest in China, 77,525 people with COVID-19 recovered.

COVID-19 is a highly contagious respiratory infectious disease that can cause respiratory, physical and psychological dysfunction in patients. Respiratory rehabilitation reduces the patient's symptoms of dyspnea, relieves anxiety and depression, reduces the patient's need to apply to the hospital, increases functional capacity and improves the patient's quality of life. Respiratory rehabilitation, according to the feedback from China, is very important for patients in the clinical treatment and recovery process after treatment. Rehabilitation of people with mild disease after discharge is mainly based on improving physical fitness and psychological adaptation. It is also aimed to gradually restore the individual's ability to the activity before the disease and return to the community as soon as possible. Individuals with COVID-19 who have respiratory and / or limb dysfunction and chronic disease after discharge should receive respiratory rehabilitation therapy. According to the current findings of the patients discharged from severe acute respiratory syndrome (SARS-CoV) and Middle East respiratory syndrome (MERS) and the clinical experience of patients with Acute Respiratory Distress Syndrome (ARDS) patients who recovered after discharge, COVID-19 patients may have physical fitness, dyspnea after activity, and muscle atrophy. (Including respiratory muscles and trunk muscles) It is recommended to use respiratory videos and booklets as the main method for respiratory rehabilitation in isolated patients at home. Telerehabilitation method is also a different recommendation option for rehabilitation.

The purpose of this study is to investigate the effects of exercises performed by telerehabilitation in patients diagnosed with COVID-19 followed at home. It is aimed to use an innovative model based on the digitally supported, home-based exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with COVID-19,
* Having been diagnosed in the last 1 week,
* Being between the ages of 18-70,
* Patients who continue to be followed at home

Exclusion Criteria:

* Hospitalization patients
* Having a serious cognitive impairment
* Having serious hearing and vision problems

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 2 weeks
  Visual Analogue Scale (VAS) is a horizontal line, 100 mm in length, and anchored by word descriptors at each end. The VAS dyspnea score uses "no shortness of breath at all" and "maximum shortness of breath" . The patient marks on the line the point that they feel represents the perception of their current state. The distance (mm) between the beginning of the horizontal line and this mark represents the degree of dyspnea perception
Modified Borg Scale | 2 weeks
  This scale used was a modified Borg scale of perceived exertion adapted to be appropriate for measuring fatigue. This consisted of a vertical scale labelled 0-10, with corresponding verbal expressions of progressively increasing perceived sensation intensity. (0 = no fatigue , 10 = maximal fatigue)
Leicester Cough Questionnaire | 2 weeks
  Leicester Cough Questionnaire (LCQ) is an English-born self-reporting quality of life measure of chronic cough. It consists of 19 items with a 7 point likert response scale (range from 1 to 7). Each item is developed to assess symptoms during cough and impact of cough on three main domains: physical, psychological and social. Scores are calculated as a mean of each domain and the total score is calculated by adding every domain score. It generally takes about 5 minutes to be completed and it is designed for adults
Timed Up and Go | 2 weeks
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance.
  It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. During the test, the person is expected to wear their regular footwear and use any mobility aids that they would normally require
30 Second Chair Stand Test | 2 weeks
  The 30-s Chair Stand Test consists of standing up and sitting down from a chair as many times as possible within 30 seconds. A standard chair without backrest, but with armrests is used. Initially, the person is seated on the chair with his backs upright. They are told to look forward with their arms folded in their chest and rise at their preferred speed after the command "1, 2, 3, go". All trials must be carried out using the same chair and similar environmental conditions.
The Beck Depression Inventory | 2 weeks
  The Beck Depression Inventory (BDI) is a 21-item, self-rated scale that evaluates key symptoms of depression. Individual scale items are scored on a 4-point continuum (0=least, 3=most), with a total summed score range of 0-63. Higher scores indicate greater depressive severity. Two subscales include a cognitive-affective subscale and a somatic-performance subscale
The Beck Anxiety Inventory | 2 weeks
  The Beck Anxiety Inventory (BAI) is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in children and adults.The questions used in this measure ask about common symptoms of anxiety . It is designed for individuals who are of 17 years of age or older and takes 5 to 10 minutes to complete. Several studies have found the Beck Anxiety Inventory to be an accurate measure of anxiety symptoms in children and adults

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No